CLINICAL TRIAL: NCT02731807
Title: A Pharmacokinetic And Relative Bioavailability Of Different Formulation Of Nutritional Supplement TA-65 In Healthy Volunteers: A Pilot, Replicate Cross-Over Study
Brief Title: TA-65 Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 15-00834
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: TA-65; Telemorase; Dietary Supplement
MeSH Terms: interventions — Powders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose A, B, C, D, E (Experimental): All participants will receive all doses throughout the course of the study.
  Interventions: Dietary Supplement: Dose A: TA-65 24mg, powder; Dietary Supplement: Dose B: TA-65, 8mg, powder; Dietary Supplement: Dose C: TA-65 3.2mg, capsule; Dietary Supplement: Dose D: TA-65 8mg, capsule; Dietary Supplement: Dose E: TA-65 32mg, capsule
- Dose D, E, C, B, A (Experimental): All participants will receive all doses throughout the course of the study.
  Interventions: Dietary Supplement: Dose A: TA-65 24mg, powder; Dietary Supplement: Dose B: TA-65, 8mg, powder; Dietary Supplement: Dose C: TA-65 3.2mg, capsule; Dietary Supplement: Dose D: TA-65 8mg, capsule; Dietary Supplement: Dose E: TA-65 32mg, capsule
- Dose C, D, E, A, B (Experimental): All participants will receive all doses throughout the course of the study.
  Interventions: Dietary Supplement: Dose A: TA-65 24mg, powder; Dietary Supplement: Dose B: TA-65, 8mg, powder; Dietary Supplement: Dose C: TA-65 3.2mg, capsule; Dietary Supplement: Dose D: TA-65 8mg, capsule; Dietary Supplement: Dose E: TA-65 32mg, capsule
- Dose E, D, C, B, A (Experimental): All participants will receive all doses throughout the course of the study.
  Interventions: Dietary Supplement: Dose A: TA-65 24mg, powder; Dietary Supplement: Dose B: TA-65, 8mg, powder; Dietary Supplement: Dose C: TA-65 3.2mg, capsule; Dietary Supplement: Dose D: TA-65 8mg, capsule; Dietary Supplement: Dose E: TA-65 32mg, capsule

INTERVENTIONS:
Dietary Supplement: Dose A: TA-65 24mg, powder
  Other Names: CAG
Dietary Supplement: Dose B: TA-65, 8mg, powder
Dietary Supplement: Dose C: TA-65 3.2mg, capsule
Dietary Supplement: Dose D: TA-65 8mg, capsule
Dietary Supplement: Dose E: TA-65 32mg, capsule

SUMMARY:
This study is a pilot research study in humans to determine the steady state pharmacokinetic profile of TA-65 after oral dose of formulated and unformulated forms. There will be eight (8) subjects of healthy men and women (non-child bearing). TA-65 is supposed to supplement the diet to increase general health through telomerase activation.The active ingredient in TA-65 activates an enzyme called telomerase. However, the active ingredient has poor oral bioavailability in humans. This study is created to enhance the bioavailability in telomerase with different formulations; powder and capsule form.

DETAILED DESCRIPTION:
This is an open labeled, replicate cross-over study with eight (8) subjects which will include men and women (non childbearing age) and be completed over a period of six (6) weeks. The supplement TA-65 will be given to subjects in both capsules and powder form.

TA-65 is a dietary supplement. The active ingredient is isolated from roots of Astragalus species. The active ingredient has been proven to activate an enzyme called telomerase. TA-65 in intended to supplement the diet to increase the general health through telomerase activation. The active ingredient has poor oral bioavailability in humans. The current study is aimed at assessing the bioavailability of the active ingredient with different formulations designed to enhance the bioavailability.

The objective of the study is to determine the steady state pharmacokinetic profile of TA-65 following oral dose of formulated (powder and capsules) and unformulated (powder) forms as assessed by Cmax, Tmax and AUC (area under the curve).

This will be a pilot, open-label, replicate cross-over study to evaluate the pharmacokinetic profile of active ingredient in eight subjects following the oral intake of TA-65 varying in formulations and doses. The subjects are expected to participate in this study for a period of 28 days. After initial screening, all subjects will visit the study center on five different days (day 1, day 7, day 14, day 21 and day 28). During each visit, all eight subjects will orally take one of the five test materials.

The washout period is seven days during which all subjects refrain from taking TA-65 in any form.

Pharmacokinetic sampling for measurement of plasma concentrations will be conducted over a 12 hour period following the oral dose. Blood will be withdrawn from all subjects prior to the intake of the test materials (0 hr.) and 1, 2, 3, 4, 5, 7, 10 and 12 hours following the oral intake of the test material. Serum will be separated from each blood sample and stored at -20° C. The amount of TA-65 in each serum samples will be analyzed by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or non-childbearing potential females, 22-55 years of age
* Subjects who have signed a written informed consent consistent.
* BMI ≥ 18.5 and ≤ 32.0 at screening with a maximum weight of 120 kg
* Medically healthy and good health as deemed by PI
* Subjects who are not on any medication or dietary supplement.
* Subjects who are able to follow the protocol as designed by TA Science and NYU

Exclusion Criteria:

* History of serious medical condition or psychiatric condition
* Subject is mentally or legally incapacitated or has significant emotional problems at the time of screening visit
* Recent history of myocardial infarction.
* Subjects with a history of cancer within the last 5 years.
* Subjects currently taking any prescribed medications or any OTC (over-the-counter) dietary supplements.
* History of drug or alcohol addiction.
* Females who are pregnant, lactating, or nursing or who may become pregnant during the course of the study.
* Patients diagnosed as HIV-positive, diagnosed with AIDS.
* Clinically significant infection within 3 months prior to screening as determined by the PI
* Consumption of grapefruit or grapefruit juice within seven days prior to the first dose of study medication and throughout the pharmacokinetic phase of the study.
* Patients with any condition not previously named that, in the opinion of the investigators or intake staff, would jeopardize the safety of the patient or affect the validity of the data collected in this study.
* Has donated blood within 3 months of screening visit or plans to donate blood within 3 months of study completion.
* Plasma donation within 7 days prior to dosing of test product
* Participation in another clinical trial within 30 days prior to screening.
* Allergy to heparin

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration (c max) of TA-65 in serum | 12 hours
Time to reach maximum concentration (T max) of TA-65 in serum | 12 hours
Area Under the Curve (AUC) | 12 hours
  For a given time interval (t2-t1), the AUC is calculated as follows:
  AUC =1/2 (C1+C2)(t2-t1) Where the C1 and C2 are the amount of the test product in blood at time 1 (t1) and time 2 (t2) respectively. Average concentration of test material in the body over the total time interval will be calculate by the sum of all of the intervals together from the first time point to the last.

CONTACTS AND LOCATIONS:
Overall Officials: David Keefe, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States